CLINICAL TRIAL: NCT05658185
Title: Migraine Difficult to Treat: the Importance of Psychological Care in the Chronic Patient
Acronym: MIDITRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, M. Antonia Pérez-Marín, PhD in Psychology, University of Valencia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIDITRA
Record Dates: First submitted 2022-11-01; First posted 2022-12-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2022-12

CONDITIONS: Migraine Disorders; Headache, Migraine
Keywords: Intervention study; psychopathology; coping illness; protective factors; risk factors
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Control Group (No Intervention): All patients will be evaluated on 4 occasions: 1) T1: 1st pre-treatment measurement in control and experimental groups; 2) after 10 weeks, T2: 2nd pre-treatment measurement in control and experimental groups; 3) after 10 weeks, T3: 3rd pre-treatment measurement in control and experimental groups, and 1st post-treatment measurement in experimental groups. Between T2 and T3 the patients in the experimental group will receive for 10 weeks the 10 sessions of the psychological treatment protocol; 4) after that, in the following 10 weeks, the control group will receive the 10 sessions of psychological treatment, thus at T4: 1st post-treatment measurement in the control group, and 1st post-treatment follow-up session in the experimental group (during this time, the experimental group does not receive any more treatment sessions, but practices all the psychological management skills installed during the treatment protocol between T2 and T3).
- Experimental Group (Experimental): All patients will be evaluated on 4 occasions: 1) T1: 1st pre-treatment measurement in control and experimental groups; 2) after 10 weeks, T2: 2nd pre-treatment measurement in control and experimental groups; 3) after 10 weeks, T3: 3rd pre-treatment measurement in control and experimental groups, and 1st post-treatment measurement in experimental groups. Between T2 and T3 the patients in the experimental group will receive for 10 weeks the 10 sessions of the psychological treatment protocol; 4) after that, in the following 10 weeks, the control group will receive the 10 sessions of psychological treatment, thus at T4: 1st post-treatment measurement in the control group, and 1st post-treatment follow-up session in the experimental group (during this time, the experimental group does not receive any more treatment sessions, but practices all the psychological management skills installed during the treatment protocol between T2 and T3).
  Interventions: Behavioral: MIDITRA

INTERVENTIONS:
Behavioral: MIDITRA — The psychological treatment protocol will be implemented over 10 group sessions of face-to-face psychological treatment with patients. The treatment sessions will have the following objectives and themes:
  * Adjustment to the disease:
  * Self-esteem/self-concept:
  * Coping with fear:
  * Emotional self-regulation:
  * Social area and enjoyment:
  * Decision making and problem solving:
  * Communication and listening skills:
  Arms: Experimental Group

SUMMARY:
In the study of migraine headaches, it is important to consider the affectation presented by those patients whose migraines do not respond easily to treatment. These difficult to treat patients are more likely to develop chronic headache, facilitating the appearance of psychological problems associated with this disease. Holistic care of these patients includes: the disability caused by pain, the impact of pain on their lives, the level of pain catastrophizing, perceived psychological well-being, quality of life and emotional distress. The quality of life of these patients is often severely affected and the psychoemotional symptoms are significantly elevated. The psychological impact associated with these difficult-to-treat chronic migraine patients is a neglected issue in current mental health care. Investigators propose to design a protocol for the evaluation and psychological treatment of these patients, based on cognitive-behavioral theory. After that, the psychological treatment of 10 group sessions will be implemented in a pilot sample. It will have 4 evaluation moments to be able to quantify, by means of questionnaires, the progress of the patients in the different stages of the study. The aim is to achieve an increase in the quality of life and a decrease in the interference of migraines in the patients' lives.

DETAILED DESCRIPTION:
Chronic diseases (CD) are characterized by their long duration, unpredictable changes in their course, in the person's appearance, limitations in physical capacity, prolonged dependence on medical specialists, continuous treatments and need for assistance.

Migraine is a neurological disorder characterized by episodic and recurrent attacks, which usually present with headache usually associated with hypersensitivity to external stimuli (visual, auditory, olfactory and cutaneous), nausea and vomiting. Migraine can be considered as a chronic process. Within this category, CM is diagnosed in persons in whom migraine attacks appear at least 15 days per month in the last three months, and in whom the headache and associated symptoms correspond to migraine attacks on at least 8 days per month. They are then said to suffer from chronic migraine CM. CM is considered to be the result of an increase in headache frequency over months or years, in a process called migraine transformation or chronification. CM usually affects people of productive age, causes great individual and social costs, and is associated with numerous comorbidities. Its usual treatment includes control measures to avoid migraine triggers, modification of risk factors and administration of pharmacological and non-pharmacological treatments, which both address and prevent attacks.

The prevalence of migraine in Western countries is between 10-16%, with a predominance in women of 2-3/18 (more than double in women). According to the WHO, migraine affects 6% of men and 18% of women and is the sixth most disabling disease in the world, taking into account the quality of life lost during the episodes, which in the most severe cases can involve constant pain for more than 15 days a month. These extremes affect one man for every eight women. This fact is one of the reasons why the disease has been stigmatized for so long. Evolutionarily, 2.5-3% of patients with episodic migraine (EM) develop CM annually.

These data point to the importance of knowing which factors can increase the risk of chronification and aggravation of the migraine patient. Knowing these factors allows us to better understand the mechanisms involved in the perpetuation of pain, so that investigators can act on them to modify the course of migraine and improve the quality of life of these patients. The risk factors related to these patients have been divided into three groups10-14: non-modifiable, modifiable and other factors.

Among the risk factors for chronification and aggravation in migraine patients, investigators would like to point out those that the literature indicates as modifiable, highlighting significantly the impact of aspects such as: stressful life events, sleep disorders, degree of disability caused by migraines, impact of the headache on daily life, level of catastrophizing about the pain, perception of psychological well-being, perceived quality of life and level of existing emotional distress (anxiety, depression, stress).

It is often difficult to treat patients with CM pharmacologically and obtain satisfactory results for them. Within the existing medical therapeutic possibilities, it is necessary to help the patient to form real expectations of the efficacy and safety of each treatment, as well as the possibilities they offer to control their disease. In this regard, there are very few studies in the scientific literature that apply psychological care protocols in this particular type of chronic patients (with CM) with clinical symptoms resistant to improvement. There is research related to chronic pain in other types of clinical conditions (back pain, pain associated with neoplasms...), but it is very scarce in patients with chronic resistant migraine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic migraine difficult to treat for at least 6 months.
* Be of legal age
* Sign the informed consent form

Exclusion Criteria:

* Failure to meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-29 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change Emotional Distress Baseline T1, Baseline T2-Pre, Post-Treatment T3 and Follow-up T4. | T1. Start T2.10 weeks after T1, T3. Evaluation 10 weeks after T2, after the intervention is finished. T4. Follow-up, 10 weeks after post-treatment.
  Assessment with Hospital Anxiety and Depression Scale in caregivers (HADS): Screening instrument for the detection of affective disorders, in non-psychiatric subjects who go to hospitals. The scale is made up of 14 items, with a range of scores from 0 to 42. The interpretation is that the higher the score, the greater the presence of anxiety-depressive symptoms.
Change in Perception of psychological stress. Baseline T1, Baseline T2-Pre, Post-Treatment T3 and Follow-up T4. | T1. Start T2.10 weeks after T1, T3. Evaluation 10 weeks after T2, after the intervention is finished. T4. Follow-up, 10 weeks after post-treatment.
  Assessment with EEP-10. The Spanish version of the EEP-10 used by Remor in a validation study with adults in Spain was used. The scale includes a series of direct queries that explore the level of stress experienced during the last month. The items are easily understood. The scale provides five response options: 'never', 'hardly ever', 'occasionally', 'many times' and 'always', which are ranked from zero to four.
Change in quality of life. Baseline T1, Baseline T2-Pre, Post-Treatment T3 and Follow-up T4. | T1. Start T2.10 weeks after T1, T3. Evaluation 10 weeks after T2, after the intervention is finished. T4. Follow-up, 10 weeks after post-treatment.
  Assessment with MSQ 21. (Migraine-Specific Quality of Life Questionnaire or MSQ)21 is a migraine-specific questionnaire designed to assess limitations in quality of life and the effect of treatments.

SECONDARY OUTCOMES:
Change in Disability due to migraine headaches. Baseline T1, Baseline T2-Pre, Post-Treatment T3 and Follow-up T4. | T1. Assessment CG and EG; T2.After 10 weeks, assessment CG and EG; T3. After 10 weeks,EG follow-up and CG evaluation after program implementation assessment after intervention application in EG; T4: follow-up evaluation in experimental and post-treatment
  MIDAS scale. This questionnaire is used to define the loss of days in all personal, professional and family areas during the last 3 months due to migraine attacks. In addition, the questionnaire allows to classify the degree of disability in null or minimal, mild, moderate and severe.
Change in Negative impact of headache. Baseline T1, Baseline T2-Pre, Post-Treatment T3 and Follow-up T4. | T1. Assessment CG and EG; T2.After 10 weeks, assessment CG and EG; T3. After 10 weeks,EG follow-up and CG evaluation after program implementation assessment after intervention application in EG; T4: follow-up evaluation in experimental and post-treatment
  The Headache Impact Test (HIT) is a tool used to measure the impact headaches have on your ability to function at work, home, school and in social situations.
  school and in social situations. Your score shows you the effect headaches have on normal daily life and your ability to function.
  It also has cut-off points that allow you to determine the degree of impact, from no impact, some impact, major impact and severe impact.
Change in Catastrophizing to pain. Baseline T1, Baseline T2-Pre, Post-Treatment T3 and Follow-up T4. | T1. Start T2.10 weeks after T1, T3. Evaluation 10 weeks after T2, after the intervention is finished. T4. Follow-up, 10 weeks after post-treatment.
  The PCS is a 13-item self-administered scale and one of the most widely used to one of the most widely used scales to assess pain catastrophism.
  In it, subjects refer to their past painful experiences and indicate the degree to which they experienced each of the 13 thoughts or feelings on a 5-point Likert scale ranging from 0 (never) to 4 (never). 5-point Likert scale ranging from 0 (never) to 4 (always).
  A total score is obtained from the scale reflecting the level of catastrophism in the face of the level of catastrophism in the face of the subject's pain. It comprises rumination, magnification and despair. The theoretical range of the instrument is between 13 and 62, with low scores indicating low catastrophizing, and high values indicating high catastrophizing.
Change in Life Satisfaction Baseline T1, Baseline T2-Pre, Post-Treatment T3 and Follow-up T4. | T1. Start T2.10 weeks after T1, T3. Evaluation 10 weeks after T2, after the intervention is finished. T4. Follow-up, 10 weeks after post-treatment.
  SWLS is a questionnaire consisting of 5 questions, with each question providing a score between 1 and 7. The maximum possible score is therefore 35. Higher scores indicate higher life satisfaction.
Change in Positive and negative affect. Baseline T1, Baseline T2-Pre, Post-Treatment T3 and Follow-up T4. | T1. Start T2.10 weeks after T1, T3. Evaluation 10 weeks after T2, after the intervention is finished. T4. Follow-up, 10 weeks after post-treatment.
  The PANAS or Positive Affect and Negative Affect Affect Scale is a self-report questionnaire. The list is divided into two segments or mood scales. One scale measures a person's positive emotion and the other scale measures negative emotion. Each segment has ten terms, which can be rated on a scale of 1 to 5 to indicate the extent to which the respondent accepts that this applies to him/her.
Change in Resilience. Baseline T1, Baseline T2-Pre, Post-Treatment T3 and Follow-up T4. | T1. Start T2.10 weeks after T1, T3. Evaluation 10 weeks after T2, after the intervention is finished. T4. Follow-up, 10 weeks after post-treatment.
  Connor-Davidson Resilience Scale to assess the ability to cope with stress and adversity. The resilience scale is made up of 10 items, with a range of scores from 0 to 40, with higher scores indicating greater resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Marián Pérez-Marín, PhD, Principal Investigator — Universitat de Valencia
Locations (2):
- Spain (2):
  - Marián Pérez-Marín, Valencia, Valencia
  - Marián Pérez-Marín, Valencia

IPD SHARING:
Plan to Share IPD: No
The database may be requested from the principal investigator upon reasonable request.